CLINICAL TRIAL: NCT06814210
Title: CAP-TEER: CerebrAl Protection During Transcatheter Edge-to-edge Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiao-dong Zhuang (Other)
Responsible Party: Sponsor-Investigator, Xiao-dong Zhuang, Dr., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAP-TEER
Record Dates: First submitted 2025-01-19; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Mitral Regurgitation; Functional Mitral Regurgitation; Degenerative Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebral Embolic Protection (Experimental): Subjects will undergo M-TEER following placement of the cerebral embolic protection device.
  Interventions: Device: Cerebral Embolic Protection
- Control Arm (No Intervention): Subjects will undergo M-TEER without cerebral embolic protection device.

INTERVENTIONS:
Device: Cerebral Embolic Protection — Subjects will undergo M-TEER following placement of the cerebral embolic protection device.
  Arms: Cerebral Embolic Protection

SUMMARY:
Transcatheter edge-to-edge repair of the mitral valve (M-TEER) is a well-established endovascular treatment option for patients with severe mitral regurgitation who are at high risk for surgery-related complications. However, the procedure carries a risk of clinically overt strokes and imaging-detected brain lesions, which may potentially be mitigated through the use of cerebral protection devices.

This prospective, multi-center, randomized, controlled study aims to assess the efficacy and safety of cerebral protection device, compared to a control group undergoing unprotected M-TEER.

DETAILED DESCRIPTION:
Subjects with indications for M-TEER and who meet study eligibility criteria will be randomized 1:1 to one of two treatment arms: 1) intervention: cerebral protection device with M-TEER or 2) Control: Unprotected M-TEER.

Enrolled subjects will undergo a diffusion weighted magnetic resonance imaging (DW-MRI) at baseline and at 72 hours, to evaluate any new cerebral lesions. Enrolled subjects will be followed for 30 days.

The study aims to address:

* To determine whether the total amounts of new brain lesion assessed by diffusion weighted magnetic resonance images at 72 hours is comparable between the experimental group and the control group.
* To assess the effectiveness and safety of cerebral protection device in the prevention of perioperative cerebrovascular events after M-TEER
* To explore the correlation between the volume/number/location of new brain lesions and changes in neurocognitive function
* To evaluate the histopathological features of the captured fragments and their relevance to clinical features

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following criteria:

General Inclusion Criteria

* Age ≥18 years
* Severe Mitral Regurgitation (3+ to 4+)
* Symptom status: NYHA functional class ≥ II
* Subjects scheduled to receive the M-TEER per the current approved indications for use
* Subjects agreed to join the study and complete follow-up

Exclusion Criteria:

Potential Subjects will be excluded if ANY of the following criteria apply:

General Exclusion Criteria

* Contraindication to MRI
* CABG, PCI, TAVR, CRT or CRT-D within the prior 30 days
* Aortic or tricuspid valve disease requiring surgery or transcatheter intervention
* COPD requiring continuous home oxygen therapy or chronic outpatient oral steroid use
* Cerebrovascular accident within prior 30 days
* Severe symptomatic carotid stenosis (>70% by ultrasound)
* Carotid surgery or stenting within prior 30 days
* Hemodynamic instability requiring inotropic support or mechanical heart assistance
* Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months.
* Contraindication for transesophageal echocardiography
* Life expectancy < 1 year
* Pregnant or planning pregnancy within next 12 months
* Participation in another interventional Trial
* Patients who are not able to give consent or complete the follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Total amounts of new lesions | 72 hours
  Total amounts of new lesions in the brain assessed by diffusion weighted magnetic resonance imaging (DW-MRI) at 72 hours.

SECONDARY OUTCOMES:
Total new lesion volume | 72 hours
  Total new lesion volume assessed by diffusion weighted magnetic resonance imaging (DW-MRI) at 72 hours
Incidence of delirium | 7 days
  Incidence of delirium
NIHSS worsening | 30 days
  NIHSS worsening
Incidence of peri- and postprocedural stroke | 30 days
  Incidence of peri- and postprocedural stroke
Incidences of MACCE at 30 days | 30 days and 1 year
  The incidences of Major Adverse Cardiac and Cerebrovascular Events (MACCE) at 30 days defined as all-cause mortality, all stroke, life-threatening or disabling bleeding, major vascular complications, and acute kidney injury (stage 2 or 3, including renal replacement therapy)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No